CLINICAL TRIAL: NCT00542659
Title: Plasma ANP and NT-pro-BNP, Atrial Anatomical Change May Determine the Outcome of Maze Operation
Brief Title: Biochemical Marker to Predict the Recurrence of Atrial Fibrillation After Surgical Maze Procedure
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Young Keun On, MD, Samsung Medical Center
Other Study IDs: 2005-02-019
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Maze procedure
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma mRNA
Oversight: Data Monitoring Committee: No

SUMMARY:
The role of plasma NT-proBNP, hsCRP, TIMP-1(Tissue inhibitors of MetalloProteinase-1),TGF-b, MMP-3(Matrix MetalloProteinase-3), and pro-MMP-1 in predicting the recurrence of AF after surgical Maze procedure.

The association of expression of CTGF, TGF-b, BNP, ANP, collagen-1, and collagen-3 in LA with the recurrence of AF after surgical Maze procedure.

ELIGIBILITY:
Inclusion Criteria:

* The patients who have valvular heart disease with atrial fibrillation and are scheduled for operation

Exclusion Criteria:

* Coronary heart disease
* Congestive heart failure

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who have valvular heart disease with atrial fibrillation and are scheduled for operation
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2005-02; Primary Completion 2007-12 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
AF recurrence | year

CONTACTS AND LOCATIONS:
Overall Officials: Young Keun On, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea